CLINICAL TRIAL: NCT00003799
Title: Phase I Study of Preoperative Radiation Therapy With Concurrent Protracted Continuous Infusion 5-FU and Dose Escalating Oxaliplatin Followed by Surgery, 5-FU, and Leucovorin for Locally Advanced (T3 and T4) Rectal Adenocarcinoma
Brief Title: Chemotherapy, Radiation Therapy, and Surgery in Treating Patients With Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03145; E1297; U10CA021115 (NIH); CDR0000066943 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Rectum; Mucinous Adenocarcinoma of the Rectum; Signet Ring Adenocarcinoma of the Rectum; Stage IIA Rectal Cancer; Stage IIB Rectal Cancer; Stage IIC Rectal Cancer; Stage IIIA Rectal Cancer; Stage IIIB Rectal Cancer; Stage IIIC Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Fluorouracil; Oxaliplatin; Radiotherapy; Radiation; Leucovorin

ARMS (1):
- Treatment (chemotherapy, radiotherapy, surgery) (Experimental): Patients receive fluorouracil IV continuously with concurrent radiotherapy for 5.5 weeks. Patients also receive oxaliplatin IV over 2 hours on day 1 of weeks 1, 3, and 5.
  Patients undergo surgery 6-8 weeks after completing preoperative chemotherapy and radiotherapy. The surgical procedure is determined by the extent of the tumor before preoperative therapy. The type of operative procedure may be abdominoperineal resection, low anterior resection (LAR), or LAR/coloanal anastomosis.
  Postoperative chemotherapy begins within 6 weeks after surgery, comprising leucovorin calcium and fluorouracil IV on days 1-5. Treatment repeats every 21 days for 4 courses.
  Interventions: Drug: fluorouracil; Drug: oxaliplatin; Radiation: radiation therapy; Drug: leucovorin calcium; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Procedure: therapeutic conventional surgery — Undergo surgery

SUMMARY:
Phase I trial to study the effectiveness of radiation therapy plus chemotherapy followed by surgery and additional chemotherapy in treating patients who have advanced nonmetastatic primary cancer of the rectum. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy, radiation therapy, and surgery may be an effective treatment for rectal cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify maximally tolerated dose (MTD) and dose limiting toxicity (DLT) of oxaliplatin when combined preoperatively with concurrent radiation therapy (XRT) and fluorouracil (5-FU) by PVI.

II. To evaluate the resection rate for T4 rectal cancers, the pathologic CR rate for T3 and T4 rectal cancers, and the expected versus actual type of resection (APR vs. LAR vs. LAR/coloanal anastomosis).

III. To make preliminary observations of patient survival and patterns of recurrence for this treatment combination.

IV. To evaluate anastomotic and sphincter function following pre-op combined modality therapy.

OUTLINE: This is a dose-escalation study of preoperative oxaliplatin.

Patients receive fluorouracil IV continuously with concurrent radiotherapy for 5.5 weeks. Patients also receive oxaliplatin IV over 2 hours on day 1 of weeks 1, 3, and 5.

Cohorts of 5 patients each receive escalating doses of oxaliplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 5 patients experience dose-limiting toxicity. Additional patients are treated at the MTD.

Patients undergo surgery 6-8 weeks after completing preoperative chemotherapy and radiotherapy. The surgical procedure is determined by the extent of the tumor before preoperative therapy. The type of operative procedure may be abdominoperineal resection, low anterior resection (LAR), or LAR/coloanal anastomosis.

Postoperative chemotherapy begins within 6 weeks after surgery, comprising leucovorin calcium and fluorouracil IV on days 1-5. Treatment repeats every 21 days for 4 courses.

Patients are followed every 3 months for 2.5 years, every 6 months for 3 years, then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, locally advanced, non-metastatic primary T3 or T4 primary adenocarcinoma of the rectum
* No evidence of tumor outside of the pelvis including liver metastases, peritoneal seeding, or metastatic inguinal lymphadenopathy
* No intra-operative radiotherapy (IORT) or brachytherapy will be allowed
* The distal border of the tumor must be at or below the peritoneal reflection, defined as within 12 centimeters of anal verge by proctoscopic examination
* Transmural penetration of tumor through the muscularis propria must be demonstrated by either of the following:

  * CT scan plus endorectal ultrasound or
  * MRI
* Tumors must be defined prospectively by the surgeon as clinically resectable or not; clinically resectable tumors will be defined by the surgeon as mobile and completely resectable with negative margins based on the routine examination of the non-anesthetized patient; before pre-op treatment, the surgeon should estimate and record the type of resection anticipated: APR, LAR, or LAR/coloanal anastomosis
* The tumor may be clinically fixed or initially not completely resectable, clinical stage T4, N0-2, M0 based on the presence of at least one of the following criteria:

  * Clinically fixed tumors on rectal examination with tumor adherent to the pelvic sidewall or sacrum
  * Sciatica attributed to sacral root invasion with CT scan/MRI evidence of the lack of clear tissue plane will be considered evidence of fixation
  * Hydronephrosis on CT scan or IVP or ureteric or bladder invasion as documented by cystoscopy and cytology or biopsy, or invasion into prostate
  * Vaginal or uterine involvement
* ECOG performance status 0-2 and surgical evaluation confirms the patient's medical condition would tolerate the proposed surgical procedure
* Caloric intake should be >= 1500 kilocalories/d
* WBC >= 3500/uL
* Platelets >= 100,000/uL
* Serum creatinine =< 2.0 mg/dL
* Serum bilirubin less than 2.0 mg/dL
* Alk Phos =< 2 x ULN
* SGOT =< 2 x ULN
* CEA should be determined prior to initiation of therapy
* Absence of clinical evidence of high-grade (lumen diameter < 1cm) large bowel obstruction, unless diverting colostomy has been performed
* Pregnant or lactating women are not eligible
* Women of childbearing potential and sexually active males are strongly advised to use an accepted and effective method of contraception
* No prior chemotherapy or pelvic irradiation therapy
* No previous or concurrent malignancy is allowed, except:

  * Nonmelanoma skin cancer or in situ cervical cancer
  * Treated non-pelvic cancer from which the patient has been continuously disease free more than five years
* No active inflammatory bowel disease or other serious medical illness which might limit the ability of the patient to receive protocol therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 1999-05; Primary Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
MTD of oxaliplatin when combined with radiation therapy and fluorouracil based on the incidence of DLT as assessed by CTC version 2.0 | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Haller, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States